CLINICAL TRIAL: NCT05353920
Title: The Effect of Cognitive Function Training Program for Community Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Huie-Ling Chiu (Other)
Responsible Party: Sponsor-Investigator, Huie-Ling Chiu, Dr., Taipei Medical University
Organization: Taipei Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: N201704031
Record Dates: First submitted 2017-12-14; First posted 2022-04-29 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-04

CONDITIONS: Cognitive Function 1, Social
MeSH Terms: interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive traiinig (Experimental)
  Interventions: Other: Cognitive training
- Active control (Active Comparator)
  Interventions: Other: Cognitive training

INTERVENTIONS:
Other: Cognitive training — cognitive related training bu virtual reality system

SUMMARY:
Background. Recently, cognitive function training program has been shown to improve cognitive function in elders. However, the effects of cognitive function training program on elderly living in the community have not been thoroughly evaluated.

Objective. The purpose of this study is to construct and evaluate the effects of cognitive function training program on cognitive function for community elderly.

Design. This is a randomized controlled study. Study subjects are elderly living in community. Subjects will be randomized into experimental group or active control group. The evaluation of the program will be evaluated at baseline, immediate after, 3 months, 6 months, and 1 year after the last session. The primary outcome indicators of the training is cognitive function, assessed by MMSE and MoCA.

Expected contribution. With rigorous design and long term follow-up, the effectiveness of cognitive function training program in Chinese population in Taiwan can be evaluated. Results of the current study will determine the value of the cognitive function training program and provide valuable information for future utilization of this protocol.

ELIGIBILITY:
Inclusion Criteria:

* 65 years old

Exclusion Criteria:

* TBI

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 62 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-08 (Actual)

PRIMARY OUTCOMES:
MMSE | 12 weeks
  cognitive function
MoCA | 12 weeks
  cognitive function

CONTACTS AND LOCATIONS:
Overall Officials: Kuei-ru Chou, Principal Investigator — Professor
Locations (1):
- TMU, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided